CLINICAL TRIAL: NCT00687180
Title: Mycophenolate vs Azathioprin in Autoimmune Hepatitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Bent Hansen, Chief of Dept. of Hepatology A-2121, Rigshospitalet, Denmark
Purpose: Treatment
Other Study IDs: MMF vs Imurel
Record Dates: First submitted 2008-05-28; First posted 2008-05-30 (Estimated); Last update posted 2008-05-30 (Estimated); Status verified 2008-05

CONDITIONS: Autoimmune Hepatitis
Keywords: Prednisolone dosage
MeSH Terms: conditions — Hepatitis, Autoimmune | interventions — Therapeutics

ARMS (2):
- I (Active Comparator): MMF
  Interventions: Drug: Treatment with mycophenolat mofetil
- II (Active Comparator)
  Interventions: Drug: Treatment with azathioprin

INTERVENTIONS:
Drug: Treatment with mycophenolat mofetil
  Arms: I
Drug: Treatment with azathioprin
  Arms: II

SUMMARY:
A study with 20 de novo patients with autoimmune hepatitis, 10 receiving azathioprin and 10 receiving mycophenolat mofetil.

ELIGIBILITY:
Inclusion Criteria:

* De novo autoimmune hepatitis
* Consent

Exclusion Criteria:

* age below 18
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet, Dept. of Hepatology A-2121, Copenhagen, Denmark